CLINICAL TRIAL: NCT03017469
Title: Achieving Resilience in Acute Care Nurses (ARISE): A Randomized Controlled Trial of a Multi-component Intervention for Nurses in Critical Care and Trauma.
Brief Title: Achieving Resilience in Acute Care Nurses (ARISE).
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Principal Investigator, Orla Smith, Director, Nursing/Clinical research, research manager, Critical Care Department, and associate scientist at the Li Ka Shing Knowledge Institute, Unity Health Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SMH30Dec2016
Record Dates: First submitted 2017-01-09; First posted 2017-01-11 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Stress, Psychological; Compassion Fatigue
Keywords: Resilience; Workplace Stress; Occupational Fatigue; Compassion Fatigue; Peer Support; Self-Care; Employee Assistance
MeSH Terms: conditions — Stress, Psychological; Compassion Fatigue; Occupational Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARISE Intervention (Experimental): Nurses who participate in the 1.5 day ARISE Intervention
  Interventions: Other: ARISE
- Control Group (No Intervention): Nurses who do not participate in the ARISE Intervention

INTERVENTIONS:
Other: ARISE — 1. Full day (7.5 hours) workshop consisting of a resilience-focused seminar facilitated by our Employee Assistance Provider (EAP) [Shepell], an introduction to hospital based resources including EAP and health and wellness offerings, and an introduction to self-care and self-care techniques including yoga and stretches, stress relief using the senses and mindfulness
  2. Half day (3.75 hours) workshop focusing on the following self-care techniques: mindfulness, yoga and stretching, and creative and reflective reading and writing
  3. Peer support through social media engagement (closed Facebook group) for 3 months post-intervention participation
  4. Five online, instructor-guided mindfulness sessions (Zoom)
  Arms: ARISE Intervention

SUMMARY:
Nurses are exposed to myriad stressors, both in the workplace and in their everyday lives, which can lead to adverse personal and professional outcomes. While workplace stress cannot be eliminated, nurses can learn techniques to build resilience, mitigate stress, and decrease fatigue. Organizational employee health, wellness, and assistance programs are all intentioned to provide this type of support; however, nurses often lack awareness of options and opportunities, and access can be a challenge. The purpose of the proposed study is to assess the outcomes of a multi-modal intervention and toolkit, ARISE, designed to enhance resilience and promote awareness of organizational resources for health, wellness, and employee assistance. We will evaluate the impact of participation in ARISE on resilience and other outcomes in nurses in critical care and trauma settings. As a Best Practice Spotlight Organization designated by the Registered Nurses Association of Ontario (RNAO), this project will incorporate relevant recommendations from Best Practice Guidelines (BPG) related to Workplace Health, Safety, and Well-being of the Nurse; and Preventing and Mitigating Nurse Fatigue in Health Care.

ELIGIBILITY:
Inclusion Criteria:

* Nurse in the medical-surgical and trauma-neurosurgical intensive care units (MSICU and TNICU) and the medical/surgical floor (9CCN),
* full-time or part-time employment status,
* approval of clinical leader manager (CLM),
* receipt of written informed consent.

Exclusion Crieria:

* casual employment status
* inability to attend intervention days

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-10-15 (Actual)

PRIMARY OUTCOMES:
Connor Davidson Resilience Scale (CD-RISC) | 1 month post intervention

SECONDARY OUTCOMES:
Connor Davidson Resilience Scale (CD-RISC) | 3 months post intervention
Occupational fatigue and recovery (OFER) scale | 1 month post intervention
  Acute fatigue and inter-shift recovery scales only
Occupational fatigue and recovery (OFER) scale | 3 months post intervention
  Acute fatigue and inter-shift recovery scales only
Professional Quality of Life (ProQOL5) scale | 1 month post intervention
Professional Quality of Life (ProQOL5) scale | 3 months post intervention
Perceived Stress Scale (PSS) | 1 month post intervention
Perceived Stress Scale (PSS) | 3 months post intervention
Occupational Coping Self-Efficacy Questionnaire for Nurses (OCSE-N). | 1 month post intervention
Occupational Coping Self-Efficacy Questionnaire for Nurses (OCSE-N). | 3 months post intervention
Mindfulness Attention Awareness Scale (MASS) | 1 month post intervention
Mindfulness Attention Awareness Scale (MASS) | 3 months post intervention
  Mindfulness attention awareness will be measured using the Mindfulness Attention Awareness Scale (MASS).
Program Evaluation Outcomes for ARISE participants | 1 month post intervention
  For each component of the intervention, and for the ARISE program as a whole, we will ask participants to rate utility, satisfaction, and frequency of use of intervention components.
Program Evaluation Outcomes for ARISE participants | 3 months post intervention
  For each component of the intervention, and for the ARISE program as a whole, we will ask participants to rate utility, satisfaction, and frequency of use of intervention components.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aiken LH, Clarke SP, Sloane DM; International Hospital Outcomes Research Consortium. Hospital staffing, organization, and quality of care: cross-national findings. Int J Qual Health Care. 2002 Feb;14(1):5-13. doi: 10.1093/intqhc/14.1.5. PMID 11871630
- [Background] Akgum S, Al-Assaf AF, & Bakar C. Reducing Burnout among Hospital Professionals. Journal of Employee Assistance, 3:15-17, 2008.
- [Background] Alexander GK, Rollins K, Walker D, Wong L, Pennings J. Yoga for Self-Care and Burnout Prevention Among Nurses. Workplace Health Saf. 2015 Oct;63(10):462-70; quiz 471. doi: 10.1177/2165079915596102. PMID 26419795
- [Background] Brown KW, Ryan RM. The benefits of being present: mindfulness and its role in psychological well-being. J Pers Soc Psychol. 2003 Apr;84(4):822-48. doi: 10.1037/0022-3514.84.4.822. PMID 12703651
- [Background] Campbell-Sills L, Stein MB. Psychometric analysis and refinement of the Connor-davidson Resilience Scale (CD-RISC): Validation of a 10-item measure of resilience. J Trauma Stress. 2007 Dec;20(6):1019-28. doi: 10.1002/jts.20271. PMID 18157881
- [Background] Peter E, Storch JL; Canadian Nurses Association. The CNA code of ethics for registered nurses. Nurs Leadersh (Tor Ont). 2008;21(2):28-33. doi: 10.12927/cjnl.2008.19872. No abstract available. PMID 18536542
- [Background] Casella E, Mills J, Usher K. Social media and nursing practice: changing the balance between the social and technical aspects of work. Collegian. 2014;21(2):121-6. doi: 10.1016/j.colegn.2014.03.005. PMID 25109210
- [Background] Chana N, Kennedy P, Chessell ZJ. Nursing staffs' emotional well-being and caring behaviours. J Clin Nurs. 2015 Oct;24(19-20):2835-48. doi: 10.1111/jocn.12891. Epub 2015 Jul 16. PMID 26178012
- [Background] Charney DS. Psychobiological mechanisms of resilience and vulnerability: implications for successful adaptation to extreme stress. Am J Psychiatry. 2004 Feb;161(2):195-216. doi: 10.1176/appi.ajp.161.2.195. PMID 14754765
- [Background] Coetzee SK, Klopper HC. Compassion fatigue within nursing practice: a concept analysis. Nurs Health Sci. 2010 Jun;12(2):235-43. doi: 10.1111/j.1442-2018.2010.00526.x. PMID 20602697
- [Background] Connor KM, Davidson JR. Development of a new resilience scale: the Connor-Davidson Resilience Scale (CD-RISC). Depress Anxiety. 2003;18(2):76-82. doi: 10.1002/da.10113. PMID 12964174
- [Background] Craigie M, Slatyer S, Hegney DG, Osseiran-Moisson R, Gentry E, Davis S., . . . Rees C. A Pilot Evaluation of a Mindful Self-care and Resiliency (MSCR) Intervention for Nurses. Mindfulness, 7(3), 764-774, 2016. doi:10.1007/s12671-016-0516-x
- [Background] Deible S, Fioravanti M, Tarantino B, Cohen S. Implementation of an integrative coping and resiliency program for nurses. Glob Adv Health Med. 2015 Jan;4(1):28-33. doi: 10.7453/gahmj.2014.057. PMID 25694849
- [Background] Dolan G, Strodl E, Hamernik E. Why renal nurses cope so well with their workplace stressors. J Ren Care. 2012 Dec;38(4):222-32. doi: 10.1111/j.1755-6686.2012.00319.x. Epub 2012 Aug 30. PMID 22934929
- [Background] Drury V, Craigie M, Francis K, Aoun S, Hegney DG. Compassion satisfaction, compassion fatigue, anxiety, depression and stress in registered nurses in Australia: phase 2 results. J Nurs Manag. 2014 May;22(4):519-31. doi: 10.1111/jonm.12168. PMID 24926496
- [Background] Fang R, Li X. A regular yoga intervention for staff nurse sleep quality and work stress: a randomised controlled trial. J Clin Nurs. 2015 Dec;24(23-24):3374-9. doi: 10.1111/jocn.12983. Epub 2015 Oct 19. PMID 26478577
- [Background] Gauthier T, Meyer RM, Grefe D, Gold JI. An on-the-job mindfulness-based intervention for pediatric ICU nurses: a pilot. J Pediatr Nurs. 2015 Mar-Apr;30(2):402-9. doi: 10.1016/j.pedn.2014.10.005. Epub 2014 Oct 20. PMID 25450445
- [Background] Gillespie BM, Chaboyer W, Wallis M. The influence of personal characteristics on the resilience of operating room nurses: a predictor study. Int J Nurs Stud. 2009 Jul;46(7):968-76. doi: 10.1016/j.ijnurstu.2007.08.006. Epub 2007 Oct 3. PMID 17915223
- [Background] Hall LH, Johnson J, Watt I, Tsipa A, O'Connor DB. Healthcare Staff Wellbeing, Burnout, and Patient Safety: A Systematic Review. PLoS One. 2016 Jul 8;11(7):e0159015. doi: 10.1371/journal.pone.0159015. eCollection 2016. PMID 27391946
- [Background] Hart PL, Brannan JD, De Chesnay M. Resilience in nurses: an integrative review. J Nurs Manag. 2014 Sep;22(6):720-34. doi: 10.1111/j.1365-2834.2012.01485.x. Epub 2012 Nov 2. PMID 25208943
- [Background] Hegney DG, Craigie M, Hemsworth D, Osseiran-Moisson R, Aoun S, Francis K, Drury V. Compassion satisfaction, compassion fatigue, anxiety, depression and stress in registered nurses in Australia: study 1 results. J Nurs Manag. 2014 May;22(4):506-18. doi: 10.1111/jonm.12160. Epub 2013 Nov 1. PMID 24175955
- [Background] Houck D. Helping nurses cope with grief and compassion fatigue: an educational intervention. Clin J Oncol Nurs. 2014 Aug;18(4):454-8. doi: 10.1188/14.CJON.454-458. PMID 25095300
- [Background] Jackson D, Firtko A, Edenborough M. Personal resilience as a strategy for surviving and thriving in the face of workplace adversity: a literature review. J Adv Nurs. 2007 Oct;60(1):1-9. doi: 10.1111/j.1365-2648.2007.04412.x. PMID 17824934
- [Background] Kemper K, Bulla S, Krueger D, Ott MJ, McCool JA, Gardiner P. Nurses' experiences, expectations, and preferences for mind-body practices to reduce stress. BMC Complement Altern Med. 2011 Apr 11;11:26. doi: 10.1186/1472-6882-11-26. PMID 21481259
- [Background] Kemper KJ. Brief Online Mindfulness Training: Immediate Impact. J Evid Based Complementary Altern Med. 2017 Jan;22(1):75-80. doi: 10.1177/2156587216639199. Epub 2016 Mar 21. PMID 27002136
- [Background] Kemper KJ, Khirallah M. Acute Effects of Online Mind-Body Skills Training on Resilience, Mindfulness, and Empathy. J Evid Based Complementary Altern Med. 2015 Oct;20(4):247-53. doi: 10.1177/2156587215575816. Epub 2015 Mar 17. PMID 25783980
- [Background] Kemper KJ, Mo X, Khayat R. Are Mindfulness and Self-Compassion Associated with Sleep and Resilience in Health Professionals? J Altern Complement Med. 2015 Aug;21(8):496-503. doi: 10.1089/acm.2014.0281. Epub 2015 Jun 2. PMID 26218885
- [Background] Klatt M, Steinberg B, Duchemin AM. Mindfulness in Motion (MIM): An Onsite Mindfulness Based Intervention (MBI) for Chronically High Stress Work Environments to Increase Resiliency and Work Engagement. J Vis Exp. 2015 Jul 1;(101):e52359. doi: 10.3791/52359. PMID 26168365
- [Background] Klatt M, Steinberg B, Marks D & Duchemin A. Changes in physiological and psychological markers of stress in hospital personnel after a low-dose mindfulness-based worksite intervention. BMC Complementary and Alternative Medicine(12), 2014. doi:1472-6882/12/S1/O16
- [Background] Kornhaber RA, Wilson A. Enduring feelings of powerlessness as a burns nurse: a descriptive phenomenological inquiry. Contemp Nurse. 2011 Oct;39(2):172-9. doi: 10.5172/conu.2011.172. PMID 22551430
- [Background] Leners C, Sowers R, Quinn Griffin MT, Fitzpatrick JJ. Resilience and professional quality of life among military healthcare providers. Issues Ment Health Nurs. 2014 Jul;35(7):497-502. doi: 10.3109/01612840.2014.887164. PMID 24963849
- [Background] Mcdonald G, Jackson D, Vickers MH, Wilkes L. Surviving workplace adversity: a qualitative study of nurses and midwives and their strategies to increase personal resilience. J Nurs Manag. 2016 Jan;24(1):123-31. doi: 10.1111/jonm.12293. Epub 2015 Apr 13. PMID 25865519
- [Background] McDonald G, Jackson D, Wilkes L, Vickers MH. Personal resilience in nurses and midwives: effects of a work-based educational intervention. Contemp Nurse. 2013 Aug;45(1):134-43. doi: 10.5172/conu.2013.45.1.134. PMID 24099234
- [Background] Mealer M, Conrad D, Evans J, Jooste K, Solyntjes J, Rothbaum B, Moss M. Feasibility and acceptability of a resilience training program for intensive care unit nurses. Am J Crit Care. 2014 Nov;23(6):e97-105. doi: 10.4037/ajcc2014747. PMID 25362680
- [Background] Mealer M, Jones J, Moss M. A qualitative study of resilience and posttraumatic stress disorder in United States ICU nurses. Intensive Care Med. 2012 Sep;38(9):1445-51. doi: 10.1007/s00134-012-2600-6. Epub 2012 May 23. PMID 22618093
- [Background] Mealer M, Jones J, Newman J, McFann KK, Rothbaum B, Moss M. The presence of resilience is associated with a healthier psychological profile in intensive care unit (ICU) nurses: results of a national survey. Int J Nurs Stud. 2012 Mar;49(3):292-9. doi: 10.1016/j.ijnurstu.2011.09.015. Epub 2011 Oct 5. PMID 21974793
- [Background] Moorley C, Chinn T. Developing nursing leadership in social media. J Adv Nurs. 2016 Mar;72(3):514-20. doi: 10.1111/jan.12870. Epub 2016 Jan 6. PMID 26732537
- [Background] Moorley CR, Chinn T. Nursing and Twitter: creating an online community using hashtags. Collegian. 2014;21(2):103-9. doi: 10.1016/j.colegn.2014.03.003. PMID 25109208
- [Background] Moss M, Good VS, Gozal D, Kleinpell R, Sessler CN. An Official Critical Care Societies Collaborative Statement: Burnout Syndrome in Critical Care Health Care Professionals: A Call for Action. Am J Crit Care. 2016 Jul;25(4):368-76. doi: 10.4037/ajcc2016133. PMID 27369038
- [Background] Sun N, Lv DM, Man J, Wang XY, Cheng Q, Fang HL, Fu Z, Liu S, Wu QH. The correlation between quality of life and social support in female nurses. J Clin Nurs. 2017 Apr;26(7-8):1005-1010. doi: 10.1111/jocn.13393. PMID 27219501
- [Background] Panagioti M, Panagopoulou E, Bower P, Lewith G, Kontopantelis E, Chew-Graham C, Dawson S, van Marwijk H, Geraghty K, Esmail A. Controlled Interventions to Reduce Burnout in Physicians: A Systematic Review and Meta-analysis. JAMA Intern Med. 2017 Feb 1;177(2):195-205. doi: 10.1001/jamainternmed.2016.7674. PMID 27918798
- [Background] Pisanti R, Lombardo C, Lucidi F, Lazzari D, Bertini M. Development and validation of a brief Occupational Coping Self-Efficacy Questionnaire for Nurses. J Adv Nurs. 2008 Apr;62(2):238-47. doi: 10.1111/j.1365-2648.2007.04582.x. PMID 18394036
- [Background] Potter P, Deshields T, Berger JA, Clarke M, Olsen S, Chen L. Evaluation of a compassion fatigue resiliency program for oncology nurses. Oncol Nurs Forum. 2013 Mar;40(2):180-7. doi: 10.1188/13.ONF.180-187. PMID 23448743
- [Background] Poulsen AA, Sharpley CF, Baumann KC, Henderson J, Poulsen MG. Evaluation of the effect of a 1-day interventional workshop on recovery from job stress for radiation therapists and oncology nurses: A randomised trial. J Med Imaging Radiat Oncol. 2015 Aug;59(4):491-498. doi: 10.1111/1754-9485.12322. Epub 2015 Jun 10. PMID 26094782
- [Background] Rushton CH, Batcheller J, Schroeder K, Donohue P. Burnout and Resilience Among Nurses Practicing in High-Intensity Settings. Am J Crit Care. 2015 Sep;24(5):412-20. doi: 10.4037/ajcc2015291. PMID 26330434
- [Background] Schmidt GB, Lelchook AM, & Martin JE.The relationship between social media co-worker connections and work-related attitudes. Computers in Human Behavior, 55: 439-445, 2016. DOI: 10.1016/j.chb.2015.09.045
- [Background] Sexton JD, Pennebaker JW, Holzmueller CG, Wu AW, Berenholtz SM, Swoboda SM, . . . Sexton JB. Care for the caregiver: benefits of expressive writing for nurses in the United States. Progress in Palliative Care, 17(6): 307-312, 2009. doi:10.1179/096992609x12455871937620
- [Background] Sheldon KM, Abad N, Hinsch C. A two-process view of Facebook use and relatedness need-satisfaction: disconnection drives use, and connection rewards it. J Pers Soc Psychol. 2011 Apr;100(4):766-75. doi: 10.1037/a0022407. PMID 21280967
- [Background] Sherrill WM, Harris M. Enhancing patient-provider communication through bibliotherapy: a brief historical review. Journal of Poetry Therapy, 27(2): 8, 2014.
- [Background] Sherring S, Knight D. An exploration of burnout among city mental health nurses. Br J Nurs. 2009 Nov 12-25;18(20):1234-40. doi: 10.12968/bjon.2009.18.20.45114. PMID 20081659
- [Background] Songprakun W, McCann TV. Evaluation of a bibliotherapy manual for reducing psychological distress in people with depression: a randomized controlled trial. J Adv Nurs. 2012 Dec;68(12):2674-84. doi: 10.1111/j.1365-2648.2012.05966.x. Epub 2012 Mar 1. PMID 22381065
- [Background] Songprakun W, McCann TV. Using bibliotherapy to assist people to recover from depression in Thailand: Relationship between resilience, depression and psychological distress. Int J Nurs Pract. 2015 Dec;21(6):716-24. doi: 10.1111/ijn.12250. Epub 2014 Mar 12. PMID 24621304
- [Background] Sorenson C, Bolick B, Wright K, Hamilton R. Understanding Compassion Fatigue in Healthcare Providers: A Review of Current Literature. J Nurs Scholarsh. 2016 Sep;48(5):456-65. doi: 10.1111/jnu.12229. Epub 2016 Jun 28. PMID 27351469
- [Background] Steege LM, Pinekenstein B. Addressing Occupational Fatigue in Nurses: A Risk Management Model for Nurse Executives. J Nurs Adm. 2016 Apr;46(4):193-200. doi: 10.1097/NNA.0000000000000325. PMID 27011153
- [Background] Wei W, Taormina RJ. A new multidimensional measure of personal resilience and its use: Chinese nurse resilience, organizational socialization and career success. Nurs Inq. 2014 Dec;21(4):346-357. doi: 10.1111/nin.12067. Epub 2014 Apr 8. PMID 24707977
- [Background] Weidlich CP, Ugarriza DN. A pilot study examining the impact of care provider support program on resiliency, coping, and compassion fatigue in military health care providers. Mil Med. 2015 Mar;180(3):290-5. doi: 10.7205/MILMED-D-14-00216. PMID 25735019
- [Background] Windle G, Bennett KM, Noyes J. A methodological review of resilience measurement scales. Health Qual Life Outcomes. 2011 Feb 4;9:8. doi: 10.1186/1477-7525-9-8. PMID 21294858
- [Background] Winwood PC, Colon R, McEwen K. A practical measure of workplace resilience: developing the resilience at work scale. J Occup Environ Med. 2013 Oct;55(10):1205-12. doi: 10.1097/JOM.0b013e3182a2a60a. PMID 24064782
- [Background] Winwood PC, Winefield AH, Dawson D, Lushington K. Development and validation of a scale to measure work-related fatigue and recovery: the Occupational Fatigue Exhaustion/Recovery Scale (OFER). J Occup Environ Med. 2005 Jun;47(6):594-606. doi: 10.1097/01.jom.0000161740.71049.c4. PMID 15951720
- [Background] Winwood PC, Winefield AH, Lushington K. Work-related fatigue and recovery: the contribution of age, domestic responsibilities and shiftwork. J Adv Nurs. 2006 Nov;56(4):438-49. doi: 10.1111/j.1365-2648.2006.04011.x. PMID 17042823
- [Background] Wittenberg-Lyles E, Goldsmith J, Reno J. Perceived benefits and challenges of an oncology nurse support group. Clin J Oncol Nurs. 2014 Aug;18(4):E71-6. doi: 10.1188/14.CJON.E71-E76. PMID 25095307
- [Background] Yates PJ, Benson EV, Harris A, Baron R. An investigation of factors supporting the psychological health of staff in a UK emergency department. Emerg Med J. 2012 Jul;29(7):533-5. doi: 10.1136/emj.2010.099630. Epub 2011 Jun 27. PMID 21708961
- See also: Registered Nurses' Association of Ontario [RNAO]. (2011). Preventing and Mitigating Nurse Fatigue in Health Care Toronto, Canada Registered Nurses' Association of Ontario — http://rnao.ca/bpg/guidelines/preventing-and-mitigating-nurse-fatigue-health-care
- See also: Stamm, B. (2005 ). The ProQOL Manual: THE PROFESSIONAL QUALITY OF LIFE SCALE: Compassion Satisfaction, Burnout & Compassion Fatigue/Secondary Trauma Scales. Pocatello, ID. — http://www.compassionfatigue.org/pages/ProQOLManualOct05.pdf